CLINICAL TRIAL: NCT03723213
Title: Investigation of Activity Daily Living Performance in Patients With Chronic Stroke
Brief Title: Activity Daily Living Performance in Patients With Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Çiğdem Çekmece, assistant professor, Kocaeli University
Other Study IDs: KU GOKAEK 2018/251
Record Dates: First submitted 2018-10-23; First posted 2018-10-29 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-10

CONDITIONS: Stroke
Keywords: stroke; occupational therapy; activity daily living
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the rehabilitation of stroke patients, the emphasis is on the treatment of physical pathologies such as increased range of motion and muscle strength, reduction of spasticity and pain. All these treatments provide increased physical capacity of the patient. But these are not enough for perform the activity daily living. In order to be successful in activity daily living of the patient, performance based treatment methods should also be applied.

The use of Canadian Occupational Performance Measurement (COPM), which measures patients' defined problem areas in daily practice should contribute to the patient-oriented approach process.

DETAILED DESCRIPTION:
In the rehabilitation of stroke patients, the emphasis is on the treatment of physical pathologies such as increased range of motion and muscle strength, reduction of spasticity and pain. All these treatments provide increased physical capacity of the patient. But these are not enough for perform the activity daily living. In order to be successful in activity daily living of the patient, performance based treatment methods should also be applied.

The use of Canadian Occupational Performance Measurement (COPM), which measures patients' defined problem areas in daily practice should contribute to the patient-oriented approach process.The Canadian Occupational Performance Measure (COPM) is an important tool to enable personalized health care.One of the strengths of the measure is its broad focus on occupational performance in all areas of life, including self-care, leisure and productivity, taking into account development throughout the lifespan and the personal life circumstances.

COPM has been described as having various advantages in terms of increasing applicability, responsibility and motivation for occupational therapy.There are two focus points in the COPM. The first one is the person-centered; the second is activity performance appropriate to the person's wishes.

By using conventional methods in stroke rehabilitation, contractures and deformities that may occur in patients can be reduced, muscle strength can be increased, and inadequate gait failure in patients can be minimized.

However, in many activities needed for daily living activities, the patient is able to sustain his inadequacy such as dressing, eating, bathing, going to the store. With the application of COPM, deficiencies in patients and the most important needs can be emphasized; thus, a program can be prepared during the treatment process. As the COPM test is a patient-centered test, it has an important place in occupational therapy programs.

In this study, Frenchay Activities Index, Barthel ADL Index and COPM will be applied in order to focus on the performances that stroke patients need in their daily living activities and to improve the independence of the patients and to emphasize patient-focused treatment. After the tests are applied, the rehabilitation process will be conducted by a treatment plan according to the needs of the patients.After the treatments, the tests will be repeated and the success rate will be evaluated on the patients.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 between 65 years of age,
* To be volunteer,
* Stability of medical conditions of patients,
* Have a sufficient communication skills,
* There will be not severe pain that will affect the treatment
* At least three months after cerebrovascular disease,
* Hemiplegia depends on cerebrovascular disease
* There will be not serious cognitive defect [Mini Mind Test (MMT) score of 24 and above],
* The patients have to have Stage of Brunnstrom is III or more appropriate,
* Modified Ashworth Scale (MAS) score has to be 2 and below
* Independent seating balance

Exclusion Criteria:

* To be an acute term stroke
* Patient consciousness is closed,
* Having a history of stroke before,
* Having a history of spinal cord lesion, traumatic brain injury, other accompanying neurological disease (multiple sclerosis, Parkinson's disease, dementia) or lower motor neuron disease,
* Having a history of tumor, convulsion,
* An important comorbid disease, such as severe heart disease (aortic stenosis, angina, arrhythmia, pacemaker) and uncontrolled hypertension, which may prevent rehabilitation, epileptic seizure history,
* No volunteer
* Excessive spasticity in the affected upper extremity joints (shoulder, elbow, wrist, fingers) [Modified Ashworth Scale (MAS) score is ≥ 3,
* Lack of sitting balance

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: In this study we will take patients depends on a article's statistics that called "Combined Cognitive-Strategy and TaskSpecific Training Improve Transfer to Untrained Activities in Subacute Stroke: An Exploratory Randomized Controlled Trial". We calculated the power analysis from this article. According to this calculated; α=0.05, 1-β=0.20, influence quantity=0.69.
  Between September 10, 2018 and February 11, 2019, 26 stroke patients between the ages of 18-65 who applied for rehabilitation treatment in Kocaeli University Faculty of Medicine Department of Physical Medicine and Rehabilitation will be included.
Sampling Method: Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2018-10-24 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2019-10-11 (Estimated)

PRIMARY OUTCOMES:
canadian occupational performance measure (COPM) | 3 weeks interval
  COPM has a client-centered design and measures outcomes according to three occupational performance areas (self-care, productivity, and leisure), examining self-perceived changes in the occupational performance of patients through a semistructured interview. The COPM prompts discussion between interviewees and therapists on factors such as different areas of activity, their concerns, and problems to be resolved. At the beginning, patients start by identifying their difficulties according to the three occupational performance areas. They subsequently use a 10-point Likert-type scale, ranging from not at all crucial (1) to extremely crucial (10), to identify the intensity of certain difficulties. For the top five problems or tasks selected by patients, the interviewer asks them to continue identifying their performance and satisfaction with their performance by using the same 10-point rating scale. Accordingly, therapists focus on these main problems or tasks.

SECONDARY OUTCOMES:
Modified Ashworth Scale (MAS) | 3 weeks interval
  The MAS measures resistance during passive soft-tissue stretching and is used as a simple measure of spasticity.
  Scoring:
  0: No increase in muscle tone
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension 1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the range of motion
  2. More marked increase in muscle tone through most of the range of motion, but affected part(s) easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension Patients will be evaluated according to the modified ashworth scale described above.
  Spasticity of patients with MAS score 2 and below does not affect daily living activities very much. MAS has a minimal spasticity in patients with a total score of 2 and below.
Brunnstrom's Hemiplegia Recovery Staging | 3 weeks interval
  Therapist evaluates patient who suffered from stroke for determine the stage of recovery.
  There are a total of six stages in the Upper Extremity Motor Recovery Phase. There are a total of six stages in the Motor Recovery Phase. In the investigator's study, 3 or more points will be accepted for each staging.
Mini Mental Stage Examination | 3 weeks interval
  The Mini Mental State Examination (MMSE) is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. It is also used to estimate the severity and progression of cognitive impairment and to follow the course of cognitive changes in an individual over time; thus making it an effective way to document an individual's response to treatment.
The Barthel Activity Daily Living Index | 3 weeks interval
  Occupational therapist evaluates each patient in activity daily living. This scale include 10 items such as feeding (score between 0 and 10), bathing (score between 0 and 5), grooming (score between 0 and 5), dressing (score 0 and 10), bowels (score beween 0 and 10), bladder (score between 0 and 10), toilet use (score between 0 and 10), transfers (score berween 0 and 15), mobility (score between 0 and 15), stairs (score between 0 and 10).
  Evaluation of total score; 0-20: fully dependent 21-61: highly dependent 62-90: moderately dependent 91-99: slightly dependent 100: fully independent Patients with a score of 90 and above had more status.
The Frenchay Activities Index (FAI) | 3 weeks interval
  FAI is a measure of instrumental activities of daily living for use with patients recovering from stroke.
  Frenchay activity index consists of 15 items. The first 10 items are evaluated in the last 3 months. Each item is awarded a score of 0-3. The first 10 items are; food preparation, washing dishes after meals, clothes washing, light housework, heavy house forward, local shopping, social situations, more than 15 minutes walking outside, hobbies, ride the car or ride the bus.
  The last 5 items are evaluated in the last 6 months. Each item is awarded a score of 0-3. The last 5 items are; travel trip or car driving, horticultural, home care, reading, profitable business.
  The benefit of the FAI is that while activities of daily living scales tend to focus on issues related to self-care and mobility.
  Total scores will be compared before and after the study.

CONTACTS AND LOCATIONS:
Overall Officials: elif ozcan, Study Chair — Kocaeli University
Locations (2):
- Turkey (Türkiye) (2):
  - Cigdem Cekmece, Kocaeli, İzmit
  - Cigdem Cekmece, Kocaeli, Yahya Kaptan

IPD SHARING:
Plan to Share IPD: No